CLINICAL TRIAL: NCT01654562
Title: A Repeated Measures Study of Simvastatin on Choroideremia: Simvastatin Intervention and Reversal in Choroideremia Patients and Age-matched Controls.
Brief Title: The Short-term Effects of Simvastatin on the Vision of Males Affected by Choroideremia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study has been terminated due to limited participant enrollment.
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CHM-STATIN
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2013-09

CONDITIONS: Choroideremia
MeSH Terms: conditions — Choroideremia | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHM (Experimental): Administration of 40mg simvastatin daily, orally for 5 weeks (4-6 weeks window), followed by 5 week (4-6 week window) washout period.
  Interventions: Drug: Simvastatin
- Age-matched controls (Active Comparator): Administration of 40mg simvastatin daily, orally for 5 weeks (4-6 weeks window), followed by 5 week (4-6 week window) washout period.
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 40mg daily by mouth for 5 weeks (4-6 week window) followed by 5 week washout period (4-6 week window).
  Other Names: Zocor

SUMMARY:
Primary objective: To examine the short-term effects of of simvastatin on the vision on males with choroideremia, evaluated by full-field scotopic threshold testing. The investigators hypothesize that they will see a reversible decrease in the dark-adapted vision in participants taking simvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Male
* Diagnosed with choroideremia and in good health
* Willing to allow his general practitioner and consultant, if appropriate, to be notified of participation in the study
* Over age of 18 years

Exclusion Criteria:

* Female
* Significant health disease, disorder, or medication, which, in the opinion of the investigator, would put the patient at risk if he were to take simvastatin
* Already taking simvastatin or another statin

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Full-field scotopic threshold | 5 weeks (4-6 weeks)
  Full-field scotopic threshold measured at 4-6 weeks after simvastatin administration.

SECONDARY OUTCOMES:
Microperimetry, OCT, fundus autofluorescence, ERG, VA | 5 weeks (4-6 weeks)
  Correlation of retinal structure and function with changes in FST after administration of simvastatin.
Microperimetry, OCT, fundus autofluorescence, ERG, VA | 5 weeks (4-6 weeks)
  Correlation of retinal structure and function with changes in FST after washout of simvastatin.
Full-field scotopic threshold | 5 weeks (4-6 weeks)
  Full-field scotopic threshold after washout of simvastatin.

CONTACTS AND LOCATIONS:
Overall Officials: Ian M MacDonald, MD, CM, Principal Investigator — University of Alberta
Locations (1):
- Ophthalmology Research Office, University of Alberta, Edmonton, Alberta, Canada